CLINICAL TRIAL: NCT06943755
Title: A Phase 2/3, Multicenter, Randomized Open-Label Study of Zanzalintinib vs Everolimus in Participants With Previously Treated, Unresectable, Locally Advanced or Metastatic Neuroendocrine Tumors
Brief Title: Zanzalintinib Versus Everolimus in Participants With Locally Advanced or Metastatic Neuroendocrine Tumors
Acronym: STELLAR-311
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL092-311; 2025-521043-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neuroendocrine Tumor (pNET); Extra-Pancreatic Neuroendocrine Tumor (epNET)
Keywords: Metastatic Cancer; Locally Advanced Cancer; Neuroendocrine Tumor (NET)
MeSH Terms: conditions — Adenoma, Islet Cell; Neoplasm Metastasis; Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zanzalintinib (Experimental): Participants will receive zanzalintinib oral tablets once daily.
  Interventions: Drug: Zanzalintinib
- Everolimus (Active Comparator): Participants will receive everolimus oral tablets once daily.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Zanzalintinib — Administered as specified in the treatment arm.
  Other Names: XL092
  Arms: Zanzalintinib
Drug: Everolimus — Administered as specified in the treatment arm.
  Other Names: Afinitor
  Arms: Everolimus

SUMMARY:
The primary purpose of this study is to assess the effectiveness of zanzalintinib compared to everolimus in participants with previously treated, unresectable, locally advanced or metastatic neuroendocrine tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed, locally advanced/unresectable or metastatic, well-differentiated Grade 1, 2, or 3 NETs of pancreatic origin or extra-pancreatic origin.
* Allowed prior lines of therapy, based on the site of NET and functional status.
* Documented radiographic disease progression per RECIST 1.1, as assessed by the Investigator based on imaging assessments (computed tomography [CT] or magnetic resonance imaging [MRI]) within 12 months before randomization.
* Measurable disease according to RECIST 1.1 as determined by the Investigator.
* Archival tumor tissue is required, if available. If archival tumor tissue is not available, a fresh biopsy may be submitted if it can be safely and feasibly obtained. Every attempt should be made to provide tumor tissue.

Key Exclusion Criteria:

* Histologically confirmed neuroendocrine carcinomas (including small cell lung cancer), medullary thyroid cancer, pheochromocytoma, paraganglioma, Merkel cell carcinoma, and mixed neuroendocrine non-neuroendocrine neoplasm (MiNEN).
* Prior treatment with a vascular endothelial growth factor receptor (VEGFR) -targeting tyrosine kinase inhibitor or a mammalian target of rapamycin (mTOR) inhibitor.
* Systemic chemotherapy and any liver-directed or other ablative therapy within 4 weeks before randomization.
* Systemic radionuclide therapy within 6 weeks before randomization.
* Radiation therapy for bone metastases within 2 weeks, any other radiation therapy, except as indicated above, within 4 weeks before randomization.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1 as Assessed by Blinded Independent Central Review (BICR) | Up to 48 months

SECONDARY OUTCOMES:
PFS Per RECIST 1.1 as Assessed by Investigator | Up to 48 months
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR and Investigator | Up to 48 months
Overall Survival (OS) | Up to 60 months
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR and Investigator | Up to 48 months
Disease Control Rate (DCR) Per RECIST 1.1 as Assessed by BICR and Investigator | Up to 48 months
Change From Baseline in Participant-Reported Global Health Status (GHS) and Disease-Related Symptoms as Assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) Score | Up to 48 months
Change From Baseline in Participant-Reported GHS and Disease-Related Symptoms as Assessed by EORTC Gastrointestinal Neuroendocrine Tumor module (QLQ-GI.NET21) Score | Up to 48 months
Number of Participants With Adverse Events | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (25):
- United States (22):
  - Exelixis Clinical Site #18, Beverly Hills, California
  - Exelixis Clinical Site #16, Los Angeles, California
  - Exelixis Clinical Site #12, Santa Monica, California
  - Exelixis Clinical Site #19, Washington D.C., District of Columbia
  - Exelixis Clinical Site #11, Tampa, Florida
  - Exelixis Clinical Site #9, Lexington, Kentucky
  - Exelixis Clinical Site #23, Metairie, Louisiana
  - Exelixis Clinical Site #8, Boston, Massachusetts
  - Exelixis Clinical Site #1, Grand Rapids, Michigan
  - Exelixis Clinical Site #5, St Louis, Missouri
  - Exelixis Clinical Site #25, Omaha, Nebraska
  - Exelixis Clinical Site #14, Albuquerque, New Mexico
  - Exelixis Clinical Site #7, New York, New York
  - Exelixis Clinical Site #17, Chapel Hill, North Carolina
  - Exelixis Clinical Site #6, Durham, North Carolina
  - Exelixis Clinical Site #20, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #21, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #24, Knoxville, Tennessee
  - Exelixis Clinical Site #10, Grapevine, Texas
  - Exelixis Clinical Site #15, Salt Lake City, Utah
  - Exelixis Clinical Site #3, Charlottesville, Virginia
  - Exelixis Clinical Site #13, Fairfax, Virginia
- Puerto Rico (2):
  - Exelixis Clinical Site #2, San Juan
  - Exelixis Clinical Site # 4, San Juan
- Exelixis Clinical Site #22, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No